CLINICAL TRIAL: NCT03702465
Title: Assessment of the Impact of a Personalised Nutrition Intervention in Impaired Glucose Regulation
Acronym: ASPIRE-DNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: DnaNudge Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18HH4629
Record Dates: First submitted 2018-10-05; First posted 2018-10-11 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Pre Diabetes
Keywords: Type 2 Diabetes; DNA-based diet; App
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Parallel assignment with an active control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Active Comparator): Pre-diabetic participants will receive general health guidelines according to the NICE guidelines, as per standard care. These will be delivered via an initial consultation with a dietitian. Participants in the control group will receive 2 follow up phone calls from the dietitian to answer any questions they may have during the study.
  Interventions: Other: Control arm
- Intervention Arm (Active Comparator): DNA-based dietary intervention: participants will receive DNA-based health guidelines via a genetic report. These will be delivered via an initial consultation with a dietitian. Participants in the control group will receive 2 follow up phone calls from the dietitian to answer any questions they may have during the study.
  Interventions: Other: DNA-based dietary intervention
- Exploratory Arm (Experimental): DNA-based dietary intervention using an app: participants will receive DNA-based health guidelines via the DnaNudge App.
  Interventions: Other: DNA-based dietary intervention using an app

INTERVENTIONS:
Other: DNA-based dietary intervention — The DNA for all arms of the study will be analysed for pre-determined single nucleotide polymorphisms (SNPs) relevant to metabolism. Participants in the intervention arm, will be provided with a hard-copy of a genetic report, which will explain how their SNPs influence their dietary habits.
  Arms: Intervention Arm
Other: DNA-based dietary intervention using an app — The DNA for all arms of the study will be analysed for pre-determined single nucleotide polymorphisms (SNPs) relevant to metabolism. Participants in the exploratory arm, will be given personalised DNA-based dietary advice via the DnaNudge App.
  Arms: Exploratory Arm
Other: Control arm — Standard care for pre-diabetic individuals: dietary advice as per the NICE guidelines for individuals who have pre-diabetes.
  Arms: Control Arm

SUMMARY:
This study will determine if DNA-based dietary guidelines can improve glucose regulation in pre-diabetic individuals significantly more than standard dietary guidelines following 6 weeks of the intervention. This will be assessed using an oral glucose tolerance test, which is a standard clinical measurement used to assess impaired glucose regulation. Pre-diabetic individuals will be recruited by offering the opportunity to self-assess their risk score for type 2 diabetes using the Leicester Risk Score Questionnaire on the Diabetes United Kingdom website, and they can contact the clinical trial team if they are interested in participating in the trial. They will then be invited for a point of care Hba1c test to determine their suitability for the trial. The point of care Hba1c test is a simple finger prick test to assess glucose regulation.

The potential for lifestyle interventions to reduce the progression to type 2 diabetes from pre-diabetic states has been demonstrated in a number of randomised control trials (RCTs) in different countries, with a meta-analysis of RCTs suggesting that lifestyle intervention in high risk subjects can halve the incidence of diabetes. However, they have been expensive and labour intensive, with multiple personal contacts. Furthermore, DNA based dietary advice has shown a greater improvement in fasting glucose measurements in obese individuals compared to standard dietary advice, with the BMI (body mass index) only showing a long-term improvement in the group that received DNA-based dietary advice. The proposed study may be able to show that increased benefits can be obtained by following a DNA-based diet compared to standard dietary advice for individuals with pre-diabetes. Furthermore, the exploratory arm of the study will receive the advice via an app (provided by DnaNudge Ltd), which if effective, would demonstrate a low-cost, widely-distributable method that could be deployed to the general public without requiring individuals to self-identify as pre-diabetic to receive an intervention.

DETAILED DESCRIPTION:
Diabetes is amongst the most common long term conditions, with the number of people affected worldwide quadrupling from 108 million in 1980 to 422 million in 2014. Its prevalence in people over 18 years of age has risen from 4.7% in 1980 to a staggering 8.5% in 2014. In 2012, there were 1.5 million deaths as a direct result of diabetes, making it the 8th leading cause of death amongst both sexes, and the 5th leading cause of death amongst women. There were a further 2.2 million deaths as a result of complications due to higher-than-optimal glucose levels. In 2013, 6% of the UK adult population (2.7 million people) were diabetic, 90% of whom had type 2 diabetes. A further 5 million people were estimated to be at high risk of developing type 2 diabetes. This has led to a cost of £8 billion per year to the NHS, 80% of which is due to diabetes-related complications such as cardiovascular disease, amputations, renal failure and sight loss.

The standard treatment protocol for pre-diabetic individuals in the UK is a brief consultation with their clinician highlighting the dangers of an increased risk of diabetes, and some general information regarding healthy eating and the benefits of regular physical activity. The individual will subsequently be contacted every 3 years to assess the state of their glucose regulation. Despite the implementation of this system, incidence rates of diabetes have continued to rise over the years. From 1994-2011, the number of women diagnosed with diabetes has risen from 1.9 - 4.9%, and 2.9 - 7.0% for men. In response to this, the NHS launched the NHS Diabetes Prevention Program (DPP) in 2016. The aforementioned studies and the predictions of the DPP are in agreement that an intensive lifestyle intervention can radically reduce incidence rates of diabetes. However, these interventions are costly, labour-intensive and require the health system to pre-identify pre-diabetic patients. The latter is one of the greatest challenges to any diabetes prevention program, as many at-risk individuals will not self-assess to pre-empt a glucose regulation test.

The investigator's solution aims to assess the improvement in glucose regulation by following a DNA-based diet in comparison with the standard protocol. The DNA-based diet will be devised based on metabolism-based genotypic traits of the participant. The traits cover metabolic imbalances such as carbohydrate sensitivity and fat sensitivity. This nutrigenetic information will be supplied to the user in an easy to use electronic format to provide food recommendations on demand during grocery shopping e.g. via the DnaNudge App or other visual indicator.

If effective, this solution could provide a cost-effective, widely-distributed, easily scalable prevention tool for improving glucose regulation in high risk individuals. Moreover, the non-invasive nature of the intervention, paired with the autonomy that it provides the individual in choosing their food choices, enables it to be a low-risk intervention. Furthermore, as a DNA-based diet is relevant for the general public, it has the potential to perform the preventative measures on individuals who do not self-identify as pre-diabetic.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Adults over 18 years of age
* Impaired glucose regulation including impaired fasting glucose (IFG) and impaired glucose tolerance (IGT) by fasting glucose, oral glucose tolerance test (OGTT) or HbA1c criteria
* Access to smart phone with an operating system of iOS 8.0 or above, or Android 4.0 or above.

Exclusion Criteria:

* Diabetic
* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Use of psychiatric, anti-diabetic, and/or weight loss medication, and/or oral steroids
* Bariatric surgery
* History of illnesses that could interfere with the interpretation of the study results (e.g. HIV, Cushing syndrome, chronic kidney disease, chronic liver disease, hyperthyroidism, hereditary fructose intolerance, alcohol or substance abuse)
* Unable to participate due to other factors, as assessed by the Chief Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in glucose regulation between the control and intervention arm | 6 weeks
  Difference in 0 minutes glucose on 75g oral glucose tolerance test between the control arm and the intervention arm.

SECONDARY OUTCOMES:
120 minutes glucose on 75g oral glucose tolerance test | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
0 minutes glucose on 75g oral glucose tolerance test | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Concentration of glycated haemoglobin in blood | 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 12 and 26 weeks.
Weight | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
BMI | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Lean mass | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Fat mass | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Waist circumference | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Measurement of total cholesterol in blood | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Measurement of fasting triglycerides in blood | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Measurement of LDL cholesterol in blood | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Measurement of HDL cholesterol in blood | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 6, 12 and 26 weeks
  Derived from measurements of insulin and glucose in blood. Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Measurement of 120 minute c-peptide | 6, 12 and 26 weeks
  Measured after a 75g oral glucose tolerance test. Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Systolic blood pressure | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Diastolic blood pressure | 6,12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Dietary intake | 6,12 and 26 weeks
  Dietary intake will be assessed using 24-hours recall questionnaire (food frequency questionnaire [FFQ]) at visits 4, 5, 7, 9 and 11. Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Energy intake from a food frequency questionnaire | 6,12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Carbohydrate intake from a food frequency questionnaire | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Fat intake from a food frequency questionnaire | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Saturated fat intake from a food frequency questionnaire | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Salt intake from a food frequency questionnaire | 6,12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Concentration of Vitamin D in blood | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Concentration of Vitamin B6 in blood | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Vitamin B12 from a food frequency questionnaire | 6, 12 and 26 weeks
  Cross-arm and within arm differences (compared to 0 week measurements) between the control arm, intervention arm, and the exploratory arm, measured at 6, 12 and 26 weeks.
Number of participant withdrawals in the trial | 26 weeks
  Number of participant withdrawals in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, M. D., Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karvela M, Golden CT, Bell N, Martin-Li S, Bedzo-Nutakor J, Bosnic N, DeBeaudrap P, de Mateo-Lopez S, Alajrami A, Qin Y, Eze M, Hon TK, Simon-Sanchez J, Sahoo R, Pearson-Stuttard J, Soon-Shiong P, Toumazou C, Oliver N. Assessment of the impact of a personalised nutrition intervention in impaired glucose regulation over 26 weeks: a randomised controlled trial. Sci Rep. 2024 Mar 5;14(1):5428. doi: 10.1038/s41598-024-55105-6. PMID 38443427
- See also: ASPIRE-DNA Clinical Trial Website — http://www.imperial.ac.uk/nudgeomics/aspire-dna-clinical-trial/

DOCUMENTS (2):
  • Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT03702465/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03702465/SAP_001.pdf